CLINICAL TRIAL: NCT04555161
Title: An Early Feasibility Study Assessing Treatment of Pulmonary Hypertension Using the Aria CV Pulmonary Hypertension System
Brief Title: Treatment of Pulmonary Arterial Hypertension Using the Aria CV Pulmonary Hypertension System
Acronym: ASPIRE PH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aria CV, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASPIREPH202001
Record Dates: First submitted 2020-08-31; First posted 2020-09-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension; Pulmonary Hypertension; Right Heart Dysfunction
Keywords: Pulmonary Disease; Pulmonary Artery; Pulmonary Hypertension; Lung Disease; Right Heart Dysfunction
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Lung Diseases

STUDY DESIGN:
Intervention Model Description: This is a single-arm, non-randomized early feasibility study to evaluate the safety and feasibility of the Aria CV PH System in patients with pulmonary hypertension and right heart dysfunction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Aria CV Pulmonary Hypertension System (Experimental): Treatment with the Aria CV Pulmonary Hypertension System
  Interventions: Device: Aria CV Pulmonary Hypertension System

INTERVENTIONS:
Device: Aria CV Pulmonary Hypertension System — The Aria CV PH System is indicated for the treatment of adult patients diagnosed with Pulmonary Hypertension in World Health Organization (WHO) Groups I, II, and III who remain symptomatic despite treatment with optimal medical therapy.
  Other Names: Aria CV PH System

SUMMARY:
This prospective study is a multi-center early feasibility study assessing the safety and performance of the Aria CV Pulmonary Hypertension System in patients with pulmonary hypertension and right heart dysfunction.

DETAILED DESCRIPTION:
This clinical investigation is a prospective, non-randomized, single-arm, multi-center early feasibility study of the Aria CV Pulmonary Hypertension (PH) System implanted in patients with pulmonary hypertension (PH). The purpose of this study is to validate that the clinical use of the Aria CV PH System is safe for the patient and to evaluate its performance in treating patients with PH and right heart dysfunction.

The study will be conducted in a maximum of 20 centers in the United States and up to 30 patients will receive implants.

Patients will be evaluated at each of the following time intervals: pre-operative, implant procedure, 7-day (or discharge if earlier), and 1-, 2-, 3-, 4-, 6-, 9-, 12-, 15-, 18-, 21-, and 24-months post index procedure. The Aria CV PH System will be assessed at each follow-up visit. The duration of the study is anticipated to last about 2 years for each patient.

ELIGIBILITY:
Common Inclusion Criteria:

1. 18 years of age or older.
2. Mean pulmonary artery pressure (mPAP) > 25mmHg.
3. Right heart dysfunction as evidence by at least one of the following:

   1. Tricuspid Annulus Plan Systolic Excursion (TAPSE) ≤ 16mm
   2. RV Fractional area change < 35%
   3. RV systolic velocity < 11.5 cm/s
   4. RV free wall strain < 18%
   5. Lateral tricuspid annulus peak systolic velocity (S') < 9cm/s
4. Pulmonary compliance (C) < 3.0 ml/mmHg
5. Current assessment of WHO FC III or ambulatory IV
6. Main pulmonary artery (MPA) diameter and anatomy suitable for placement of the device as defined in the Instructions For Use (IFU) and as assessed by multi-slice computed tomography (MSCT).
7. Subject is deemed appropriate for Aria CV device by the Subject Care Team at the investigation site and approved by the Eligibility Review Committee (ERC).
8. The subject has agreed to participate in the study by signing the study specific informed consent form.
9. The subject agrees to abide by device related travel restrictions.

   Unique Inclusion Criteria for WHO Group I:
10. Pulmonary capillary wedge pressure (PCWP) ≤ 15mmHg
11. Pulmonary vascular resistance (PVR) > 3 Woods Units (WU)
12. The subject remains symptomatic despite being on a stable drug regimen of PH specific medication(s) appropriate for their PH classification for at least 90 days prior to planned index procedure.

Unique Inclusion Criteria for WHO Group II:

10. Previous diagnosis of heart failure with preserved ejection fraction (HFpEF) (ejection fraction ≥ 50%) 11. PCWP > 15 mmHg 12. PVR > 3 WU

Unique Inclusion Criteria for WHO Group III:

10. Previous diagnosis of lung disease, including but not limited to chronic obstructive pulmonary disease (COPD) or interstitial lung disease (ILD) including idiopathic pulmonary fibrosis (IPF) or combined emphysema with fibrosis.

11. PCWP ≤ 15mmHg 12. PVR >4 WU

Common Exclusion Criteria:

1. Diagnosis of WHO Groups 4 or 5 PH.
2. Recent clinical event(s) of any of the following:

   1. Myocardial infarction or stroke within 6 months prior to the index procedure;
   2. Sustained tachyarrhythmia (documented heart rate >110/min) within 2 months prior to the index procedure;
   3. Uncontrolled, chronic atrial fibrillation.
3. Pre-existing or requirement of emergent surgery/ intervention, or implantation of prosthetic cardiac device that, in the opinion of the investigator, may interfere with Aria CV PH System placement or function.
4. Any of the following medical history or comorbidities:

   a. History of endocarditis; b. History of unprovoked Pulmonary Embolism; c. Current renal insufficiency as demonstrated by an eGFR < 30 mL/min/1.73 m2 or end stage renal disease requiring chronic dialysis; d. Current diagnosis of scleroderma associated with: i. Any history of GI bleeding or receiving iron infusions within 2 years prior to enrollment; ii. Significant skin involvement that could compromise daily activities or the ability to receive IV medications, or sclerodactyly that causes surface ulcerations, digital ulcerations, or ulcerating calcinosis lesions.

   e. History of receiving immunosuppressant therapy as follows: i. Excluded if receiving Mycophenolate mofetil within 30 days prior to enrollment, or Rituximab within 6 months prior to enrollment, or currently receiving Prednisone at a dose > 12 mg per day at time of enrollment; ii. Excluded if any immunosuppressant other than Mycophenolate mofetil, Rituximab or Prednisone, per above.

   e. Current pulmonary veno-occlusive disease (PVOD); f. Current pulmonary capillary hemangiomatosis (PCH); g. History of clinically significant patent foramen ovale (PFO) or other inter-atrial or inter-ventricular shunt; h. History of gastric antral vascular ectasia (GAVE), gastrointestinal or intracranial bleeding which, in the opinion of the investigator, will predispose subject to major bleeding events following Aria CV device placement and warfarin anticoagulation regimen; i. Active infection requiring antibiotic therapy within two (2) weeks of procedure; j. Blood dyscrasias that may, in the opinion of investigator(s), expose subject to unacceptable procedural risks such as severe or worsening leukopenia, anemia, thrombocytopenia, untreated iron deficiency or history of bleeding diathesis or coagulopathy.
5. Anatomy is not suitable for placement of Aria CV device.
6. Right heart valve regurgitation as follows:

   1. Moderate to severe (Grade 3 or 4) pulmonary valve regurgitation;
   2. Severe (Grade 4) tricuspid valve regurgitation.
7. Hypersensitivity or contraindication to:

   1. Required medications (e.g., contrast agents, warfarin, heparin) which cannot be adequately managed;
   2. Materials in device including polyurethane, silicone, nickel, and titanium.
8. Ineligible for or refuses blood transfusion.
9. Pregnant, nursing or is planning to become pregnant in the next two years.
10. Life expectancy of less than two years.
11. Currently participating in or planning to participate in other investigational study that may interfere with the outcome of this study.
12. For subject on supplemental oxygen therapy - Subject adheres to the treatment regimen that in the opinion of the physician does not increase subject's safety.
13. Previous diagnosis of cardiac amyloidosis.

Unique Exclusion Criteria for WHO Group I:

N/A

Unique Exclusion Criteria for WHO Group II:

1. Previous diagnosis of idiopathic hypertrophic subaortic stenosis (IHSS, also known as hypertrophic obstructive cardiomyopathy - HOCM).
2. Untreated severe aortic or mitral stenosis
3. Diagnosis of heart failure with reduced ejection fraction (HFrEF)
4. Previous diagnosis of nonobstructive hypertrophic cardiomyopathy.

Unique Exclusion Criteria for WHO Group III:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint is the incidence of investigational device- or procedure-related serious adverse events (SAEs). | 30 days post-implant
  The primary safety endpoint is the incidence of investigational device- or procedure-related serious adverse events through 30 days post-index procedure.

SECONDARY OUTCOMES:
Incidence of Device Implantation Success | 7 days post-implant
  Incidence of successful implantation of the Aria CV device defined as follows:
  1. Absence of investigational device or procedure-related patient death within 7 days post index procedure based on Data Safety Monitoring Board (DSMB) adjudication;
  2. Correct positioning of the Aria CV device implantable components at the targeted locations upon completion of index procedure based on imaging; and
  3. Aria CV balloon inflates and deflates responding to cyclic pressure changes in the pulmonary artery at time of index procedure, based on imaging.
Changes in World Health Organization (WHO) Functional Class | 6 months post-implant
  Changes in WHO Functional Class from baseline to 6-month.
Changes in 6-Minute Walk Distance | 6 months post-implant
  Changes in the 6-minute walk distance from baseline to 6-month.
Changes in Modified Borg Dyspnea Score (MBS) | 6 months post-implant
  Changes in MBS from baseline to 6-months. MBS is a measure of breathlessness during exercise that ranges from 0 to 10, where 0 is no breathlessness and 10 is maximal breathlessness.
Changes in biomarker N-terminal pro hormone BNP (NT-pro-BNP) | 6 months post-implant
  Change in N-terminal pro hormone BNP (NT-pro-BNP) from baseline to 6-months.
Changes in REVEAL Score | 6 months post-implant
  Changes in REVEAL Score 2.0 from baseline to 6-months. The REVEAL 2.0 is a risk calculator for PAH patients that ranges from 0 (lowest risk) to 22 (highest risk).
Changes in quality of life as measured by the Living with Pulmonary Hypertension (LPH) questionnaire score | 6-months post-implant
  Changes in quality of life from baseline to 6-months as measured by the LPH total score. The Living with Pulmonary Hypertension (LPH) questionnaire has 21 questions each scored on a 6-point scale ranging from 0 (no) to 5 (very much). The LPH total score, calculated by summing scores for the 21 individual questions, ranges from 0 (best) to 105 (worst).
Changes in quality of life as measured by the emPHasis-10 questionnaire score | 6-months post-implant
  Changes in quality of life from baseline to 6-months as measured by the emPHasis-10 questionnaire score which assesses breathlessness, fatigue, confidence and control. The total score ranges from 0 to 50 with higher scores indicating poorer quality of life.
Incidence of Serious Adverse Events | 24 months post-implant
  Safety will be evaluated by assessing the incidence of device and/or procedure related SAEs from device implant through last follow up.
Changes in pulmonary vascular resistance (PVR) | 6 months post-implant
  Changes in PVR (Woods unit) as measured by right heart catheterization from baseline to 6 months.
Changes in pulmonary artery pressures (PAPs) | 6 months post-implant
  Changes in PAPs (mmHg) as measured by right heart catheterization from baseline to 6 months.
Changes in pulmonary capillary wedge pressure (PCWP) | 6 months post-implant
  Changes in PCWP (mmHg) as measured by right heart catheterization from baseline to 6 months.
Changes in pulmonary arterial compliance | 6 months post-implant
  Changes in pulmonary arterial compliance (L/mmHg) as measured by right heart catheterization from baseline to 6 months.
Changes in cardiac output (CO) from baseline | 6 months post-implant
  Changes in cardiac output (L/Min) as measured by right heart catheterization from baseline to 6 months.
Changes in right heart function | 6 months post-implant
  Changes in right heart function as measured by echocardiographic imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Ravichandran, M.D., Principal Investigator — Ascension Health; Jim White, M.D., Ph.D., Principal Investigator — University of Rochester
Locations (12):
- United States (12):
  - University of California - San Diego, La Jolla, California
  - University of California-Los Angeles, Los Angeles, California
  - St. Vincent Health, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cornell University, New York, New York
  - University of Rochester, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio Health, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Aurora St Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vollmers K, Scandurra J, Woolley JR, Giridharan GA, Rothman AMK, Pritzker M, Weir EK, Gerges C, Lang I. Development of a Novel, Pulmonary Endovascular Device to Treat Patients With Pulmonary Hypertension. Pulm Circ. 2025 Jul 29;15(3):e70131. doi: 10.1002/pul2.70131. eCollection 2025 Jul. PMID 40741160
- See also: Information about the Aria CV Pulmonary Hypertension System — https://ariacv.com/